CLINICAL TRIAL: NCT05979311
Title: A Phase 3b, Multi-center, Randomized, Parallel-group, Open-label, Non-inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Oral Dolutegravir/Lamivudine Once-daily as a First-line Regimen Compared to Oral Bictegravir/Emtricitabine/Tenofovir Alafenamide Once Daily for Virologic Suppression and Maintenance in Antiretroviral Therapy Naive Adults Living With HIV
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of Using an Oral Once-daily 2 Drug Regimen Compared to an Oral Once-daily 3 Drug Regimen for the Treatment of Human Immunodeficiency Virus (HIV)-1 in Adults Who Have Not Previously Taken Antiretroviral Therapy
Acronym: VOGUE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 219816
Record Dates: First submitted 2023-07-19; First posted 2023-08-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: HIV; HIV Infections
Keywords: Antiretroviral-naïve; Bictegravir; Dolutegravir; Emtricitabine; Human immunodeficiency virus 1 (HIV-1); Lamivudine; Virologic suppression; Tenofovir alafenamide
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; Lamivudine; bictegravir; Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DTG/3TC (Experimental): Participants will receive FDC of DTG/3TC once daily until Week 96.
  Interventions: Drug: Dolutegravir; Drug: Lamivudine
- BIC/FTC/TAF (Active Comparator): Participants will receive BIC/FTC/TAF once daily until Week 96.
  Interventions: Drug: Bictegravir; Drug: Emtricitabine; Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Dolutegravir — Dolutegravir will be administered once daily.
  Arms: DTG/3TC
Drug: Lamivudine — Lamivudine will be administered once daily.
  Arms: DTG/3TC
Drug: Bictegravir — Bictegravir will be administered once daily.
  Arms: BIC/FTC/TAF
Drug: Emtricitabine — Emtricitabine will be administered once daily.
  Arms: BIC/FTC/TAF
Drug: Tenofovir alafenamide — Tenofovir alafenamide will be administered once daily.
  Arms: BIC/FTC/TAF

SUMMARY:
This study will compare safety, efficacy, participant reported outcomes and implementation outcomes of a fixed dose combination (FDC) of a two-drug regimen dolutegravir (DTG) plus lamivudine (3TC) and a three-drug regimen FDC of bictegravir (BIC), emtricitabine (FTC) and tenofovir alafenamide (TAF) in HIV-1 infected adult participants who have not previously received antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age >=18 years (or older, if required by local regulations) at the time of obtaining informed consent.
* An individual participant is eligible to participate if they are not pregnant (as confirmed by a negative serum human chorionic gonadotropin (hCG) test at Screening and a negative urine hCG test at Enrollment) and not lactating.
* Antiretroviral-naïve (no prior therapy with any antiretroviral agent following a diagnosis of HIV-1 infection) person living with HIV.
* Participant (or participant's legally acceptable representative [LAR]) is capable of giving written informed consent.
* Eligible participants or their LAR must sign a written Informed Consent Form before any protocol-specified assessments are conducted. Enrollment of participants who are unable to provide direct informed consent is optional and will be based on local legal/regulatory requirements and site feasibility to conduct protocol procedures.
* Participants enrolled in France must be affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding or plan to become pregnant or breastfeed during the study.
* Any evidence of a current Centers for Disease Control and Prevention (CDC) Stage 3 disease; with the exception of cutaneous Kaposi's sarcoma not requiring systemic therapy, and CD4+ count <200 cells per cubic millimeter (neither is exclusionary).
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates study participation.
* Ongoing or clinically relevant pancreatitis.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical intraepithelial neoplasia; other localized malignancies require agreement between the Investigator and the Medical Monitor for inclusion of the participant prior to enrollment.
* Participants with severe hepatic impairment (Class C) as determined by Child-Pugh classification.
* Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of liver cirrhosis with or without hepatitis viral co-infection.
* Alanine aminotransferase (ALT) >=5 times the upper limit of normal (ULN) or ALT >=3*ULN and bilirubin >=1.5*ULN (with >35% direct bilirubin).
* Participants determined by the Investigator to have a high risk of seizures, including participants with an unstable or poorly controlled seizure disorder. A participant with a prior history of seizure may be considered for enrollment if the Investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the Medical Monitor prior to enrollment.
* Participants who, in the investigator's judgment, pose a significant suicide risk. Participant's recent history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk.
* Signs and symptoms which, in the opinion of the Investigator, are suggestive of active Coronavirus disease 2019 (COVID-19) (example fever, cough) infection within 14 days prior to enrollment.
* Evidence of Hepatitis B virus (HBV) infection based on the results of central lab testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis B surface antibody (HBsAb) and HBV Deoxyribonucleic Acid (DNA) as follows:

  a. Participants positive for HBsAg are excluded; b. Participants negative for HBsAb and negative for HBsAg but positive for hepatitis B core antibody (HBcAb) may be excluded based on the following consideration: i. Exclude if HBV DNA is detected [either <Lower Limit of Quantification (LLoQ), >Upper Limit of Quantification (ULoQ) OR numerical value (i.e., between LLoQ and ULoQ)] ii. Not excluded if HBV DNA is negative, not detected
* Participants with Hepatitis C virus (HCV) co-infection at Screening are eligible only if:

  i. liver enzymes meet entry criteria; and ii. HCV disease is not anticipated to require on-study treatment with any agent(s) that have potential adverse drug-drug interactions (DDIs) with the study interventions; and iii. HCV disease has undergone appropriate work-up and is not advanced and will not require treatment prior to the primary endpoint or later visit. Additional information on participants with HCV co-infection at screening should include results from any liver biopsy, Fibroscan, ultrasound, or other fibrosis evaluation, history of cirrhosis or other decompensated liver disease, prior treatment, and timing/plan for HCV treatment.

iv. In the event that recent biopsy or imaging data is not available or inconclusive, the Fib-4 score will be used to verify eligibility

1. Fib-4 score >3.25 is exclusionary;
2. Fib-4 scores 1.45 - 3.25 requires Medical Monitor consultation.

Fibrosis 4 score Formula:

(Age * Aspartate aminotransferase [AST]) / (Platelets * (square root of ALT)

* Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment) are excluded. Participants with a false positive RPR (with negative treponemal test) or serofast RPR result (persistence of a reactive nontreponemal syphilis test despite history of adequate therapy and no evidence of re-exposure) may enroll after consultation with the Medical Monitor. Participants who completed treatment at least 7 days prior to Screening are eligible.
* Presence of any major resistance-associated mutations as defined by the International Antiviral Society-United States of America (IAS-USA) resistance guidelines to DTG, 3TC, BIC, FTC or TAF in the Screening result.
* Exposure to an experimental drug or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent (whichever is longer), prior to first dose of study treatment.
* Treatment with any of the following agents within 28 days of Screening:

  i. radiation therapy; ii. cytotoxic chemotherapeutic agents; iii. tuberculosis therapy with the exception of isoniazid (isonicotinylhydrazid, INH); iv. immunomodulators that alter immune responses such as chronic systemic corticosteroids, interleukins, or interferons.
* Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
* Treatment with any agent with documented activity against HIV-1 in vitro within 28 days of first dose of study treatment. Treatment withacyclovir/valacyclovir is permitted.
* Participants receiving any protocol-defined prohibited medication and who are unwilling or unable to switch to an alternate medication.
* Any verified Grade 4 laboratory abnormality, with the exception of Grade 4 lipid abnormalities.
* Any acute laboratory abnormality at Screening, which, in the opinion of the investigator, would preclude the participant's participation in an interventional clinical trial.
* Participant has estimated creatine clearance <30 milliliter per minute (mL/min) per 1.73 square meter using the refitted, race-neutral Chronic Kidney Disease Epidemiology Collaboration (CKD-EPIcr_R) method.
* Participants known or suspected to have acquired HIV-1 concurrent with use of Pre-exposure prophylaxis (PrEP) or Post-exposure prophylaxis (PEP) must be discussed with the Medical Monitor prior to enrollment.
* Any condition which, in the opinion of the Investigator, may interfere with the absorption, distribution, metabolism or excretion of the study drugs or render the participant unable to receive study medication.
* Any pre-existing physical or mental condition (including substance use disorder) which, in the opinion of the Investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
* Participant is currently participating in, or anticipates being selected for, any other interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2024-02-09 (Actual); Primary Completion 2026-03-24 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with plasma HIV- Ribonucleic acid (RNA) less than (<)50 copies per milliliter (c/mL) as per snapshot algorithm at Week 48 | Week 48

SECONDARY OUTCOMES:
Percentage of participants with plasma HIV-1 RNA <50 c/mL as per snapshot algorithm at Weeks 24 and 96 | Weeks 24 and 96
Percentage of participants with HIV-RNA greater than or equal to (>=)50 c/mL as per snapshot algorithm at Weeks 24, 48, and 96 | Weeks 24, 48 and 96
Change from Baseline in HIV-1 RNA at Weeks 24, 48 and 96 | Baseline (Day 1) and Weeks 24, 48 and 96
Change from Baseline in Cluster of differentiation 4 positive (CD4+) cell count at Weeks 24, 48 and 96 | Baseline (Day 1) and Weeks 24, 48 and 96
Change from Baseline in CD4/Cluster of differentiation 8 (CD8) at Weeks 24, 48 and 96 | Baseline (Day 1) and Weeks 24, 48 and 96
Number of Participants With HIV-1 Disease Progression | Weeks 24, 48 and 96
Time to virologic suppression (HIV-1 RNA <50 c/mL) from Baseline | Baseline (Day 1) and Up to Week 96
Number of participants with confirmed virologic withdrawal (CVW) | Up to Week 96
Number of Participants with treatment-emergent resistance | Up to week 96
Change from Baseline in Renal Biomarkers- estimated glomerular filtration rate at Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in Renal Biomarkers- urinary protein/creatinine at Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in renal biomarker- Serum Cystatin C at Weeks 48 and 96 (Milligrams per liter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in renal biomarker- Serum Retinol Binding Protein (RBP) at Weeks 48 and 96 (Milligrams per deciliter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in renal biomarker- Serum Beta-2 Microglobulin (B2M) at Weeks 48 and 96 (Micrograms per milliliter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in bone biomarkers- Serum Bone Specific Alkaline Phosphatase, Serum Procollagen type 1 N- Propeptide, Serum Type I Collagen C-Telopeptides and Serum Osteocalcin at Weeks 48 and 96 (Micrograms per Liter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in bone biomarkers- Serum Vitamin D at Weeks 48 and 96 (Nanomoles per Liter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline (Week 4) in Total Treatment Satisfaction Score Using HIV Treatment Satisfaction status Questionnaire (HIVTSQs) at Weeks 12, 24, 48 and 96 (Scores on a scale) | Baseline (Week 4) and Weeks 12, 24, 48 and 96
  The HIVTSQ status version (HIVTSQs) is assessing participants' satisfaction with their current treatment with a Total score ranging from 0 to 60. Higher scores indicate a greater level of satisfaction with HIV treatment. Baseline is defined as measurement value at Week 4.
Change from Baseline (Week 4) in Individual Item Scores Using HIVTSQs at Weeks12, 24, 48 and 96 (Scores on a scale) | Baseline (Week 4) and Weeks 12, 24, 48 and 96
  Individual items scores range from 0 to 6 (0=very dissatisfied, 6=very satisfied). Baseline is defined as measurement value at Week 4.
Change from Baseline (Week 4) in Domains Scores Using HIVTSQs at Weeks 12, 24, 48 and 96 (Scores on a scale) | Baseline (Week 4) and Weeks 12, 24, 48 and 96
  There are two domain scores of General Satisfaction/Clinical and Lifestyle/Ease subscales; each comprised of 5 items with possible scores of 0 to 30. The higher the score, the greater the satisfaction within the subscale. Baseline is defined as measurement value at Week 4.
Change from Baseline in bothersome symptoms using the Symptom Distress Module at Weeks 4, 12, 24, 48 and 96 (Score on a scale) | Baseline (Day 1) and Weeks 4, 12, 24, 48 and 96
  The Symptom Distress Module (SDM) is a 20-item self-reported measure that addresses the presence and perceived distress linked to symptoms commonly associated with HIV or its treatment. Symptom bother score is based on the score for each symptom present ranging from 1 (it does not bother me) to 4 (it bothers me a lot). Symptom bother score is the unweighted sum of the bother item scores for each symptom. The symptom bother score ranges from 0 (minimum bother score) to 80 (maximum bother score).
Absolute values for waist and hip circumference (Centimeters) | Up to Week 96
Absolute values for waist to hip ratio and waist to height ratio (Ratio) | Up to Week 96
Absolute values for Body weight (Kilogram) | Up to Week 96
Absolute values for systolic and diastolic blood pressure (millimeters of mercury) | Up to Week 96
Change from Baseline in Body Mass Index (kilogram per square meter) | Baseline (Day 1) and Up to Week 96
Change from Baseline in body weight greater than (>) 5 percentage (%) at Weeks 24, 48 and 96 | Baseline (Day 1) and Weeks 24, 48 and 96
Change from Baseline in total and regional (trunk and extremities) fat assessed by Dual-energy X-ray absorptiometry (DXA) at Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in total and regional (trunk and extremities) fat-free mass assessed by DXA Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in lumbar and hip bone mineral density (BMD) assessed by DXA at Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in trabecular bone score (TBS) assessed by DXA at Weeks 48 and 96 | Baseline (Day 1), Weeks 48 and 96
  Trabecular bone score (TBS) is a lumbar spine dual-energy absorptiometry texture index, which provides information on microarchitecture skeletal quality partially independent of BMD.
Change from Baseline in fasting glucose (Millimoles per Liter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in insulin (Microunits per millilliter) | Baseline (Day 1), Weeks 48 and 96
Change from Baseline in Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) at Week 48 and Week 96 | Baseline (Day 1), Week 48 and Week 96
Change from Baseline in Hemoglobin A1c [HbA1c] at Week 48 and Week 96 (Percentage of HbA1c) | Baseline (Day 1), Week 48 and Week 96
Change from Baseline in plasma lipids (total, high-density lipoprotein [HDL], and low-density lipoprotein [LDL] cholesterol, triglycerides) (Millimoles per Liter) at Week 48 and Week 96 | Baseline (Day 1), Week 48 and Week 96
Change from Baseline in QDiabetes Score at Week 48 and Week 96 (Scores on a scale) | Baseline (Day 1), Weeks 48 and 96
  QDiabetes score defines the risk (percentage) of developing type 2 Diabetes in the next ten years. The score ranges from 0-100.
Change from Baseline in Fibrosis 4 (FIB-4) Score at Week 48 and Week 96 (Scores on a scale) | Baseline (Day 1), Weeks 48 and 96
  A value of FIB-4 scores below 1.30 is considered as low risk for advanced fibrosis; value of FIB-4 over 2.67 is considered as high risk for advanced fibrosis; and FIB-4 values between 1.30 and 2.67 are considered as intermediate risk of advanced fibrosis.
Number of participants with metabolic syndrome at Weeks 48 and 96 | Weeks 48 and 96
Change from Baseline in Framingham cardiovascular risk scores at Weeks 48 and 96 (Scores on a scale) | Baseline (Day 1), Weeks 48 and 96
  Coronary heart disease (CHD) risk at 10 years in percent (%) can be calculated with the help of the Framingham Risk Score. Individuals with low risk have 10% or less CHD risk at 10 years, with intermediate risk 10-20%, and with high risk 20% or more.
Change from Baseline in Data collection on Adverse events of anti-HIV Drugs (DAD) cardiovascular risk scores at Weeks 48 and 96 (Scores on a scale) | Baseline (Day 1), Weeks 48 and 96
  Coronary heart disease (CHD) risk at 5 years in percent can be calculated with the help of the DAD Risk Score. The 5-year risk of CHD is classified as low (<1%), moderate (1 to 5%), high (5 to 10%), or very high (>10%).
Changes from Baseline in Systolic and diastolic blood pressure at Weeks 48 and 96 millimeters of mercury (mmHg) | Baseline (Day 1), Weeks 48 and 96

CONTACTS AND LOCATIONS:
Locations (51):
- Argentina (2):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
- Belgium (3):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
- GSK Investigational Site, Hvidovre, Denmark
- France (6):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
- Germany (5):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Frankfurt
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Thessaloniki
- GSK Investigational Site, Dublin, Ireland
- Israel (4):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Rehovot
  - GSK Investigational Site, Tel Aviv
- Italy (5):
  - GSK Investigational Site, Bari
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Padua
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Sassari
- Japan (3):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Mérida, Mexico
- Poland (3):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Wroclaw
- Portugal (2):
  - GSK Investigational Site, Aveiro
  - GSK Investigational Site, Porto
- Spain (8):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Elche Alicante
  - GSK Investigational Site, La Laguna-Tenerife
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Stockholm, Sweden
- Switzerland (2):
  - GSK Investigational Site, Basel
  - GSK Investigational Site, Zurich
- United Kingdom (2):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
ViiV will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf